CLINICAL TRIAL: NCT02530619
Title: A Multicenter, Open-Label, Pilot Study of Alisertib (MLN8237), a Novel Inhibitor of Aurora Kinase A, in Adult Patients With Relapsed/Refractory Acute Megakaryoblastic Leukemia or Myelofibrosis (Including Primary and Post-Essential/Post-Polycythemic Myelofibrosis)
Brief Title: Alisertib in Treating Patients With Myelofibrosis or Relapsed or Refractory Acute Megakaryoblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Millennium Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brady Stein, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15H10; NCI-2015-01219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00200682; NU 15H10 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Acute Megakaryoblastic Leukemia; Myelofibrosis; Primary Myelofibrosis
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Primary Myelofibrosis | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (alisertib) (Experimental): Patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
The purpose of this study is to evaluate the safety of alisertib and its effect, bad and/or good, on acute megakaryoblastic leukemia (AMKL) or myelofibrosis (MF). The study drug, alisertib, is an investigational drug. An investigational drug is one that has not been approved by the U.S. Food and Drug Administration (FDA). Alisertib has shown evidence in the lab that it may have an effect on a type of cell that produces platelets. This cell is called a megakaryocyte and it is known to be defective (doesn't work well) in both AMKL and MF.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety profile of alisertib in patients with acute megakaryoblastic leukemia (AMKL) and in patients with myelofibrosis (MF).

SECONDARY OBJECTIVES:

I. Determine preliminary efficacy of alisertib in both populations.

TERCIARY OBJECTIVES:

I. Describe pharmacodynamics (PD) effects of alisertib in peripheral blood and/or bone marrow samples.

II. Evaluate the relationship between biomarker expression levels and response to alisertib.

III. Evaluate reduction in splenomegaly by palpation (MF arm only). IV. Evaluate improvement in MF symptoms (MF arm only), as assessed by the Myeloproliferative Neoplasm Symptom Assessment form (MPN-SAF).

V. Assess change in bone marrow fibrosis in patients in the MF arm.

OUTLINE:

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at approximately 30 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* AMKL PATIENTS: Patients must have a confirmed diagnosis of relapsed/refractory acute megakaryoblastic leukemia (AMKL), as defined by World Health Organization (WHO) criteria
* AMKL PATIENTS: Patients must have an Eastern Cooperative Oncology Group (ECOG) status 0-2
* AMKL PATIENTS: Total bilirubin =< 1.5 x upper limit of normal (ULN)
* AMKL PATIENTS: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* AMKL PATIENTS: Creatinine < 1.5 x ULN or calculated creatinine clearance > 30 ml/min
* AMKL PATIENTS: Prothrombin time (PT) and partial thromboplastin time (PTT) =< 1.5 x ULN
* AMKL PATIENTS: Absolute neutrophil count (ANC) >= 1500/mm^3
* AMKL PATIENTS: Platelets >= 100,000/mm^3
* AMKL PATIENTS: Hemoglobin > 9 g/dL
* AMKL PATIENTS: Patients must have estimated life expectancy of 6 months or greater
* AMKL PATIENTS: Female patients of child-bearing potential (FOCBP) must have a negative serum beta-human chorionic gonadotropin (HCG) pregnancy test within 7 days prior to registration; NOTE: a FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* AMKL PATIENTS: Female patients must meet at least one of the following conditions:

  * Must be post-menopausal for at least 1 year prior to registration (not of childbearing potential)
  * Must be surgically sterilized
  * Willing to use an acceptable method of birth control (i.e. hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* AMKL PATIENTS: Male patients, even if surgically sterilized (status post-vasectomy) agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of alisertib
* AMKL PATIENTS: Patients must be able to understand and willing to sign a written informed consent
* MF PATIENTS: Patients must have a confirmed diagnosis of myelofibrosis (MF), as defined by WHO criteria
* MF PATIENTS: Patients must be intermediate I risk or beyond and meet the following:

  * In need of treatment
  * Intolerant or refractory to ruxolitinib (or other investigational Janus kinase [JAK]-inhibitors) OR unlikely to benefit from ruxolitinib
  * Ineligible for stem cell transplantation
* MF PATIENTS: Patients must have an ECOG status 0-2
* MF PATIENTS: Direct bilirubin < 1.5 x ULN
* MF PATIENTS: ALT/AST =< 2.5 x ULN
* MF PATIENTS: Creatinine < 1.5 x ULN or calculated creatinine clearance > 30 ml/min
* MF PATIENTS: PT and PTT =< 1.5 x ULN
* MF PATIENTS: ANC >= 1500/mm^3
* MF PATIENTS: Platelets >= 100,000/mm^3
* MF PATIENTS: Patients must have estimated life expectancy of 6 months or greater
* MF PATIENTS: Female patients of child-bearing potential (FOCBP) must have a negative serum beta-HCG pregnancy test within 7 days prior to registration
* MF PATIENTS: Female patients must meet at least one of the following conditions:

  * Must be post-menopausal for at least 1 year prior to registration (not of childbearing potential)
  * Must be surgically sterilized
  * Willing to use an acceptable method of birth control (i.e. hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* MF PATIENTS: Male patients, even if surgically sterilized (i.e. status post-vasectomy) agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of alisertib
* MF PATIENTS: Patients must be able to understand and willing to sign a written informed consent

Exclusion Criteria:

* Patients who have received treatment with clinically significant enzyme inducers (such as enzyme inducing antiepileptic drugs phenytoin, carbamazepine, or phenobarbital, or rifampin, rifabutin, rafapentine, or St. John's wort) within 14 days prior to registration are not eligible
* Patients who have received any investigational products, antineoplastic therapies, or radiotherapy within 14 days prior to registration are not eligible; NOTE: patients actively receiving hydroxyurea are eligible and may continue to receive hydroxyurea through cycle 1 of protocol treatment
* Patients who have received prior administration of an Aurora A kinase targeted agent (including alisertib) are not eligible
* Patients who have received corticosteroids within 7 days prior registration are not eligible, UNLESS the patient has been taking a continuous dose of no more than 15 mg/day of prednisone for at least 1 month prior; NOTE: low dose steroid use for control of nausea and vomiting will be allowed; topical steroid use and inhaled steroids are also permitted
* Patients who are candidates (eligible and willing) for standard and/or potentially curative treatments are not eligible
* Patients who have had received radiation therapy to more than 25% of the bone marrow are not eligible (whole pelvic radiation is considered to be over 25%)
* Patients who have had major surgery within one month (28 days) prior to registration are not eligible
* Patients who have had prior allogenic bone marrow or organ transplantation are not eligible
* Patients who have had grade 2 or higher diarrhea, despite optimal antidiarrheal supportive care, within 7 days prior to registration are not eligible
* Patients who have had grade 2 or higher peripheral neuropathy within 14 days prior to registration are not eligible
* Patients who have had a myocardial infarction within 6 months (24 weeks) prior to registration are not eligible
* Patients who have class III or IV heart failure (as defined by the New York Heart Association), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities are not eligible
* Patients who have known gastrointestinal (GI) disease or GI procedures which could interfere with the oral absorption or tolerance of alisertib are not eligible; examples include (but are not limited to) partial gastrectomy, history of small intestine surgery, and celiac disease
* Patients who have a known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness (such as severe chronic obstructive pulmonary disease or requirement for supplemental oxygen) are not eligible
* Patients who have a requirement for constant administration of proton pump inhibitor, histamine-2 (H2) antagonist, or pancreatic enzymes are not eligible; intermittent usage of antacids or H2 antagonists are allowed
* Patients who have a systemic infection requiring intravenous (IV) antibiotic therapy within 14 days prior to registration (or other severe infection) are not eligible
* Patients who are known human immunodeficiency virus (HIV) positive are not eligible
* Patients who are known hepatitis B surface antigen positive are not eligible
* Patients who have known or suspected active hepatitis C infections are not eligible; NOTE: patients who are hepatitis C surface antigen positive are eligible
* Female patients who are pregnant or breast feeding are not eligible
* Patients who have a severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study are not eligible
* Patients who have symptomatic central nervous system (CNS) involvement are not eligible
* Patients who have been diagnosed or treated for another malignancy within 3 years prior to registration are not eligible aside from these exceptions: completely resected basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients who are unable to swallow oral medication or are unwilling to comply with the administration requirements are not eligible
* Patients who require administration of myeloid growth factors or platelet transfusions within 14 days prior to registration are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2022-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brady Stein, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on October 09, 2015 with an accrual goal of 24 patients. The first patient started treatment July 05, 2016. The study closed to further accrual on November 02, 2017 with total accrual having been met.
Groups:
- Alisertib 50 mg BID: Patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Alisertib: Administered orally 50 mg BID on days 1-7 of each cycle; one cycle is defined as 21 days (days 8-21 will be rest days). Patients may continue to receive cycles of alisertib until progression of disease or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Period: Registered for Study
Arm/Group | Alisertib 50 mg BID
Started | 26
Registered | 26
Received 1st Dose of Alisertib | 24
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Completed 1st Cycle of Treatment
Arm/Group | Alisertib 50 mg BID
Started | 24
Completed | 24
Not Completed | 0
Period: Continued Treatment Cycles 2 Through 6
Arm/Group | Alisertib 50 mg BID
Started | 24
Completed | 14
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 4
Not completed — Lack of Efficacy | 2
Period: Continued Treatment Cycle 7+
Arm/Group | Alisertib 50 mg BID
Started | 14
Completed | 14
Not Completed | 0
Period: Follow-up Period (6 Months)
Arm/Group | Alisertib 50 mg BID
Started (3 patients are still on treatment and have not entered the follow-up period.) | 21 (Patients who received at least one dose of study drug go into follow-up.)
Completed | 10
Not Completed | 11
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Two patients were registered to the study, but never received any study drug (alisertib). These two patients are excluded from demographics.
Arm/Group | Alisertib 50 mg BID
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24
Refractory Acute Megakaryoblastic Leukemia or Myelofibrosis [Count of Participants; unit: Participants]
  Myelofibrosis | 24
  Refractory Acute Megakaryoblastic Leukemia | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Alisertib Per NCI's Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Description: Adverse events will be defined as those included in CTCAE v 4.0. The AEs that were determined to be at least possibly related to study drug and graded 3, 4, 5 are included here. Grade 1 (mild): the event causes discomfort without disruption of normal daily activities. Grade 2 (moderate): the event causes discomfort that affects normal daily activities. Grade 3 (severe): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status. Grade 4 (Life-threatening): the patient was at risk of death at the time of the event. Grade 5 (fatal): the event caused death. All patients who received at least 1 dose of alisertib were considered evaluable for this endpoint.
Time Frame: From time of treatment to 6 months post discontinuation (range of cycles attempted 1 to 29, median 7.5 cycles, 1 Cycle = 21 days)
Population: Data was collected from all patients for the primary endpoint until May 2018 when it was determined there was sufficient data collected for primary endpoint analysis and primary endpoint was determined to be met. At the time of data cut off, 7 patients remained on active treatment and range of cycles completed by patients was 1-29 (median 7.5 cycles). No further data was collected after May 2018 for primary outcome measure purposes.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 50 mg BID
Number analyzed (Participants) | 24
Participants
  Neutropenia Grade 3 | 5
  Neutropenia Grade 4 | 5
  Febrile Neutropenia Grade 3 | 1
  Lymphocytopenia Grade 3 | 9
  Thrombocytopenia Grade 3 | 5
  Thrombocytopenia Grade 4 | 2
  Anemia Grade 3 | 5
  Vertigo Grade 3 | 1
  Diarrhea Grade 3 | 1
  Alanine aminotransferase increased Grade 3 | 1
  Creatinine increased Grade 3 | 1

2. Secondary Outcome: Response to Treatment
Description: Serial blood and/or bone marrow samples will be collected at specific timepoints for each disease to determine response to alisertib treatment.
Time Frame: Baseline to up to 6 months after the last dose of treatment
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Changes in Biomarker Expression Levels
Description: To evaluate the relationship between biomarker expression levels and response. Biomarkers will include a) genes encoding key enzymes in Aurora kinase signaling, b) markers of cellular aneuploidy and apoptosis, and c) markers of megakaryocytic differentiation.
Time Frame: Baseline to up to 6 months after the last dose of treatment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Changes in MF Symptoms Assessed by the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) Score (MF Patients)
Description: To evaluate improvement in MF symptoms in the MF arm, changes in symptom scores over time will be calculated.
Time Frame: Once per cycle (1 cycle=21 days)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Pharmacodynamic Effects of Alisertib
Description: Serial blood and/or bone marrow samples will be collected at specific timepoints. Flow cytometry, colony forming assays, AURKA autophosphorylation assays, and in vitro cultures of patient specimens to assess the effect of MLN8237 on megakaryocytes and other hematopoietic cells will be measured.
Time Frame: Baseline to up to 6 months after the last dose of treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Splenomegaly by Palpation (MF Patients)
Description: To evaluate reduction in splenomegaly by palpation in the MF arm. Patients will be examined for splenomegaly by palpation once per cycle and change from baseline will be calculated over time.
Time Frame: Baseline to up to 6 months after the last dose of treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Bone Marrow Fibrosis (MF Patients)
Description: Assess change in bone marrow fibrosis in patients in the MF arm. Bone marrow will be assessed at screening and after cycle 6 in this population.
Time Frame: Screening and up to 54 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 5 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 6 months post last treatment. 1 cycle = 21 days. Serious Adverse Events (SAEs) are reported from the time of treatment initiation. The range of cycles attempted was 1-38. At the time of reporting this data, 3 patients remain on treatment.
Arm/Group | Alisertib 50 mg BID
All-Cause Mortality (participants affected / at risk) | 5/24
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg BID (N=24)
Upper Respiratory Infection - parainfluenza (Infections and infestations) | 1 — The patient also experienced fever at the time of this event.
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 1 — The patient also experienced fever, hypoxia, encephalopathy, and renal failure at the time of this event.
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Non- ST Myocardial Infarction (NSTEMI) (Cardiac disorders) | 1
pulmonary embolism (Vascular disorders) | 1 — The patient also experienced abdominal pain at the time of this event.
Anemia (Blood and lymphatic system disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1 — The patient also experienced hyponatremia at the time of this event.
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg BID (N=24)
Anemia (Blood and lymphatic system disorders) | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 3
Edema face (General disorders) | 1
Edema limbs (General disorders) | 7
Fatigue (General disorders) | 9
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 5
Bronchial infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 4
Wound complication (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 6
Creatinine increased (Investigations) | 9
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
INR increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 16
White blood cell decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 13
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 9
Thromboembolic event (Vascular disorders) | 1
Raynaud Syndrome (Blood and lymphatic system disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Systolic murmur (Cardiac disorders) | 1
cardiomegaly (Cardiac disorders) | 1
Murmur (Cardiac disorders) | 1
Decreased Hearing (Ear and labyrinth disorders) | 1
conjunctivae erythema (Eye disorders) | 1
eye bruising and edema (Eye disorders) | 1
Retinal Hemmorhage (Eye disorders) | 1
eye redness (Eye disorders) | 1
periorbital bruising (Eye disorders) | 1
Blood in stool (Gastrointestinal disorders) | 1
polydipsia (General disorders) | 1
prostatomegaly (General disorders) | 1
Popliteal fossa cysts (General disorders) | 1
Gallstones (Hepatobiliary disorders) | 1
rhinorrhea (Infections and infestations) | 1
C difficile positive (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
tinea pedis (Infections and infestations) | 1
Night Sweats (Investigations) | 1
Pain in the bone marrow site (Injury, poisoning and procedural complications) | 1
Appetite increased (Metabolism and nutrition disorders) | 1
metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Small Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mood Swings (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
renal cysts (Renal and urinary disorders) | 1
Respiratory synctial virus (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Tear (Skin and subcutaneous tissue disorders) | 1
skin nodules (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
facial hair loss (Skin and subcutaneous tissue disorders) | 1
shoulder cyst (Skin and subcutaneous tissue disorders) | 1
calcifications (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT02530619/Prot_SAP_000.pdf